CLINICAL TRIAL: NCT05203523
Title: Investigating the Effect of Cognitive Training with and Without Transcranial Alternating Current Stimulation on the Executive Brain Functions in Dementia Population
Brief Title: Investigational Dementia Treatment Study
Acronym: tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Riverview Health Centre Foundation (Other); Charis Senior Residences LP. DBA Aster Gardens (Unknown)
Responsible Party: Principal Investigator, Dr. Zahra Kazem-Moussavi, Professor, Dept. of Electrical and Computer Eng. Director Biomedical Engineering, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HS25171(B2021:089)
Record Dates: First submitted 2021-10-03; First posted 2022-01-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2022-02

CONDITIONS: Dementia, Mild
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This human research study is a crossover, placebo controlled and double-blind study. It will have two groups of subjects matched in age, and sex and cognitive level (measured by Montreal Cognitive Assessment: MoCA).
  Group 1 (G1) participants will receive active tACS simultaneously with cognitive exercises.
  Group 2 (G2) participants will receive sham tACS simultaneously with cognitive exercises.
  The volunteers who cannot tolerate application of tACS and focus on the cognitive exercises at the same time, will be enrolled in a third group (G3); they will receive only cognitive exercises with the same protocol as in G1 and G2.
  We will use only two periods design (one time crossing over).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The group assignment is known only by the study coordinator and the PI. Group assignment will be randomized into either Group 1 or Group 2 using PROC PLAN procedure of SAS randomization. The group assignment of a participant could potentially be unblinded on compassionate ground (e.g., if a participant comes from a different city for the duration of the study) or request of the participant or any emergency situation (although very rare). In that case the participant's data may be excluded from the analysis totally or depending on when this unblinding occur, half of the data might be usable for analysis (if unblinding occur during the waiting period before crossing over). The unblinding decision will be made by the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (G1) (Experimental): Participants will receive active tACS simultaneously with cognitive exercises.
  Interventions: Device: transcranial alternative current stimulation (tACS); Other: cognitive exercises
- Group 2 (G2) (Sham Comparator): Participants will receive sham tACS simultaneously with cognitive exercises.
  Interventions: Other: cognitive exercises

INTERVENTIONS:
Device: transcranial alternative current stimulation (tACS) — A light electrical current will be applied to the scalp of the participants via 2 electrodes, while the participants performs cognitive exercises with the guidance of a trained research assistant.
  Arms: Group 1 (G1)
Other: cognitive exercises — Participant will perform memory and learning games/tasks through "Mind Triggers" app on an IPad. Participants will be guided by a highly trained research assistant.

SUMMARY:
This research investigates the effect of active versus sham tACS paired with cognitive exercises in a regimen protocol of weeks, everyday. The study design is a one-time crossing over design in which participants are randomized into two groups: One group will receive active treatment for 4 weeks, then 8 weeks of no treatment followed by another 4 weeks of treatment but with sham. The other group will start with sham and end up with active treatment. The study is double-blind; thus, neither participants, nor the assessors know the group assignment.

The Intervention is applying tACS either active or sham paired with cognitive exercises (MindTriggers app games).

Note: The above study will run at both University of Manitoba (U of M) and Aster Gardens residence. However, at Aster Gardens Residence only questionnaire type of assessments will be run, while in U of M, the investigators will have three other major assessments as well. In addition, the investigators will run the assessments at the Aster Gardens Residence through online sessions.

DETAILED DESCRIPTION:
This research will investigate the effect of applying transcranial alternating current stimulation (tACS) when paired with cognitive exercises on older adults in a placebo-controlled double-blind study with statistical rigor. In addition, the investigators will investigate and explore novel technological methods not only to monitor the plausible changes due to intervention but also to predict the response of a participant to the intervention at baseline. Since most technological intervention on dementia have a demanding and costly protocol, it would be of great interest to have a reliable prediction of a participant to a treatment at baseline; that would lead to personalized optimum treatment strategy. The investigators will use Electrovestibulography (EVestG), Egocentric Spatial Assessment using our Virtual Reality Navigation (VRN) and functional near infrared spectroscopy (fNIRS) measurements and analysis to develop the monitoring and predicting technologies. EVestG is a non-invasive measure of the vestibuloacoustic system in both background (no motion) and in response to passive whole-body tilt stimuli. The investigators hypothesize there is a direct link between vestibular system deficiencies and Alzheimer's. VRN measures how people orient themselves in a non-familiar environment; the investigators hypothesize it is deteriorated significantly in Alzheimer's even at its onset. fNIRS measures oxygenated and deoxygenated blood flow to the brain and it may help to understand neuronal changes due to intervention.

ELIGIBILITY:
Inclusion Criteria:

* ability to read, write and speak English fluently

Exclusion Criteria:

* Being diagnosed with Parkinson's, Parkinsonian dementia, Huntington disease, speech significant aphasia and intellectual disability, major depression/anxiety, bipolar disorder, schizophrenia or any other major mood disorder
* Having a History of epileptic seizures or epilepsy
* Inability to adequately communicate in English
* Impaired vision or hearing severe enough to impair performance in cognitive tests
* Current substance abuse disorder
* Currently participating in another therapeutic study for dementia
* Plan to change the medication during this study's period

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Wechsler Memory Scale (WMS-IV) Older Adult Battery Score at five, eleven and sixteen weeks. | Baseline (week 0), week 5, week 11, week 16
  Cognitive and memory task that focus on 6 major memory indexes: Auditory Memory, Visual Memory, Visual Working Memory, Immediate Memory, Delayed Memory, and Recognition Memory.

SECONDARY OUTCOMES:
N-back test | Baseline (week 0), week 5, week 11, week 16
  N is a number between 1 and 4. A sequence of random shapes is presented and the participant has to tap or say if (remember) whether a presented object is a repeat of the Nth previous object. We will use this test with N=1 as for N>1 is very challenging for dementia population to perform.
Neuropsychiatric Inventory Questionnaire (NPIQ) | Baseline (week 0), week 5, week 11, week 16
  Questionnaire used to assesses neuropsychiatric symptoms and caregiver burden The score of the NPIQ is based on the presence of a specified symptom and a separate score for severity of the symptom. For presence the minimum total score is 0, maximum score is 12. For severity the minimum total score is 0, maximum is 36. Higher scores indicate the participant is exhibiting more severe changes in behaviors.
Functional Near Infrared Spectroscopy (fNIRS) | Baseline (week 0), week 5, week 11, week 16
  fNIRS is a device designed mainly for measuring the blood flow over the prefrontal cortex. Participants will perform a verbal fluency task while the fNIRS measures signals simultaneously.
Electrovestibulography (EVestG) | Baseline (week 0), week 5, week 11, week 16
  EVestG is explored as a monitoring and predictive tool for treatment efficacy, starting at baseline. If participant's ears are free of wax, blood, scarring, then they will be eligible for electrode placement and EVestG recording.
Virtual Reality Navigation (VRN) spatial orientation test | Baseline (week 0), week 5, week 11, week 16
  The VRN test will be run in non-immersive mode using a large screen and joystick in the PI's office at Riverview Health Center by one of the VRN team member (a research assistant). This program runs only on PC. Run the "rummeego.bat" file in the folder VRN V5 to run the program. Press "s" button to rotate the building. Pressing "Esc" exits that trial and goes to next.
  The VRN has two stages: 1) Localization, 2) Navigation. The second stage will be carried out only if a participant can pass the localization stage with a score >15 (basically with no consistent side error).
Speech analysis | Baseline (week 0), week 5, week 11, week 16
  During WMS-IV assessment, participants are interviewed with a chit-chat about their daily life and events. For speech assessment, we use the first few minutes of that interview as well as the spoken parts of the WMS-IV assessment, where the participant has to recall a story, will be recorded and used. This assessment is basically signal (speech) processing of the recorded audio at each assessment time and find features that could be representative of a change due to treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Aster Gardens, Edmonton, Alberta
  - Riverview Health Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobson N, Lithgow B, Jafari Jozani M, Moussavi Z. The Effect of Transcranial Alternating Current Stimulation With Cognitive Training on Executive Brain Function in Individuals With Dementia: Protocol for a Crossover Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 27;11(4):e37282. doi: 10.2196/37282. PMID 35475789